CLINICAL TRIAL: NCT00765713
Title: Sleep Apnea-hypopnea Syndrome and Ventricular Arrhythmias in Patients With Systolic Ventricular Dysfunction and Implantable Cardioverter-defibrillator. Incidence and Effect of CPAP Treatment
Brief Title: Sleep Apnea-hypopnea Syndrome (SAHS) and Ventricular Arrhythmias
Acronym: SAHS-ICD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Universitario La Paz (Other)
Collaborators: Hospital Virgen de la Salud (Other); Hospital Universitario Virgen Macarena (Other)
Responsible Party: Rafael Peinado Peinado, Hospital Universitario La Paz
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HULP PI-719
Record Dates: First submitted 2008-10-02; First posted 2008-10-03 (Estimated); Last update posted 2013-04-02 (Estimated); Status verified 2008-09

CONDITIONS: Sleep Apnea; Ventricular Arrythmias; Systolic Left Ventricle Dysfunction
Keywords: Sleep apnea; CPAP; Ventricular arrhythmias; Defibrillator therapies
MeSH Terms: conditions — Sleep Apnea Syndromes | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- CPAP (Experimental): Continuous positive airway pressure
  Interventions: Device: Nasal continuous positive airway pressure
- Conventional (No Intervention): Hygienic-dietetic recommendations

INTERVENTIONS:
Device: Nasal continuous positive airway pressure — Nocturnal
  Arms: CPAP

SUMMARY:
Hypothesis:

The CPAP treatment diminishes the effect of ventricular arrhythmias in patients with ischemic heart disease or dilated myocardiopathy, systolic ventricular disfunction and sleep apnea-hypopnea syndrome (SAHS)Objectives: To analyze the incidence of ventricular arrhythmias (premature ventricular beat, non-sustained ventricular tachycardia and sustained ventricular tachycardia) and appropriate defibrillator therapies in patients with ischemic heart disease or dilated myocardiopathy, moderate-severe left ventricular dysfunction,with an implantable cardioverter-defibrillator (ICD) and sleep apnea. To study the effect of CPAP on the cardiac arrhythmias and on the number of appropriate defibrillator therapies.

Design:

Parallel, randomized and single-blinded multicentric study to compare CPAP vs. hygienic-dietetic recommendations.

Patients with SAHS (AHI≥15) and systolic left ventricle dysfunction patients with an ICD.

Duration: 24 months.

DETAILED DESCRIPTION:
Secondary objectives:

To compare the prevalence of SAHS in patients with ischemic heart disease or dilated myocardiopathy and moderate-severe left ventricle dysfunction with ICD with that of the general population. To study the incidence of supraventricular arrhythmias (atrial fibrillation, atrial flutter or supraventricular tachycardia) and inappropriate defibrillator therapies in these patients. To value the effect of the treatment with CPAP on the above mentioned arrhythmias. To relate the effect of ventricular and supraventricular arrhythmias with sleep parameters, cardiovascular biomarkers, inflammation and oxidative stress. To evaluate the long-term effect of the CPAP on systemic biomarkers in patients with ischemic heart disease or dilated myocardiopathy and moderate-severe left ventricle dysfunction. To evaluate the long-term effect of CPAP on the quality of life in these patients.

Sample size:

224 patients with ischemic heart disease or dilated myocardiopathy and moderate-severe left ventricle dysfunction with ICD will be included to randomize 19 SAHS subjects for arm.

ELIGIBILITY:
Inclusion Criteria:

* Previous diagnostic of ischaemic heart disease of dilated myocardiopathy
* Ejection fraction of left ventricle < 40%
* Patients with implantable cardioverter-defibrillator

Exclusion Criteria:

* Diurnal hypersomnolence with EES > 16
* Morbid obesity (BMI > 35 Kg/m2).
* Moderate-severe chronic obstructive pulmonary disease (FEV1/FVC < 70 % and FEV1 < 80 % of reference).
* Known thyroid disease.
* Previous treatment with CPAP.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 224 (Actual)
Dates: Start 2008-10; Primary Completion 2012-10 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Number of appropriate defibrillator therapies | 24 months

SECONDARY OUTCOMES:
AHI, incidence of premature ventricular beats and non-sustained ventricular tachycardia. Plasmatic levels of C-reactive protein, homocystein, pro-BNP, sTNFαR-I, IL-1b, IL-2, IL-6, IL-8, IL-8 and 8-isoprostane | 24 moths

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Garcia-Rio, PhD, Study Director — Hospital Universitario La Paz
Locations (3):
- Spain (3):
  - Hospital Universitario La Paz, Madrid, Madrid
  - Hospital Universitario Virgen de la Macarena, Seville, Sevilla
  - Hospital Virgen de la Salud, Toledo, Toledo